CLINICAL TRIAL: NCT03062137
Title: Optimal Location of Saturation Measurement During Flexible Fiberoptic Bronchoscopy
Brief Title: Finding the Optimal Location for Saturation Measurement During Flexible Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of Pulmonary Institute, Rabin Medical Center
Other Study IDs: RMC17001ctl
Record Dates: First submitted 2017-01-31; First posted 2017-02-23 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Lung Diseases; Desaturation of Blood
Keywords: bronchoscopy; saturation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: blood gas sampling

SUMMARY:
An observational comparison of different locations of saturation measurements during Flexible Bronchoscopy

DETAILED DESCRIPTION:
The study group will include 100 patients undergoing flexible fiberoptic bronchoscopy (FFB).

The patients will receive sedation with Midazolam, Fentanyl and Propofol. All patients will receive supplemental oxygen via nasal cannula (2-4 L/min) before the beginning of the procedure.

In all cases, patients will be monitored using continuous electrocardiography, pulse oximetry (on patients finger), and transcutaneous carbon dioxide and saturation (on patients earlobe), and automated noninvasive blood pressure recordings every 5 minutes. All parameters will be recorded from accepting patient to bed of procedure until 10 minutes after removal of FFB from nasopharynx.

The saturation will be measured in 3 different locations (one pulse is added in other earlobe). additionally, A blood gas sample will be taken during discrepancy between different measurements.

Immediately after the end of procedure, the measurements from 3 different monitors will be printed, and the blood sample be taken to a gas sample machine by the investigator.

Desaturation value and time will be compared between the different locations. The blood arterial saturation will be compared to other measurements taken at the same time.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 patients, adults, undergoing Flexible Fiberoptic Bronchoscopy under sedation
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Value changes between locations | Through completion of bronchoscopy procedure an average of 30 minutes
  Difference of 10% of blood saturation between different locations during sedation for bronchoscopy procedure.
Time changes between locations | Through completion of bronchoscopy procedure an average of 30 minutes
  The level of desaturation of 90% is checked in the different monitors and the gap in seconds is registered

SECONDARY OUTCOMES:
gap between arterial gas sample and different monitors | Through completion of bronchoscopy procedure an average of 30 minutes
  during differences of more than 5% between finger and earlobe monitors we will take an arterial blood sample and the lab result will be compared to the measurements at the same time

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Principal Investigator — Rabin Medical Center, Belinson Hospital
Locations (1):
- Pulmonary Institute Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No